CLINICAL TRIAL: NCT01221792
Title: A Randomized, Double-Blind, Placebo-Controlled, Flexible-Dose Study to Assess the Safety and Efficacy of Carvedilol Versus Placebo in the Treatment of Post Traumatic Stress Disorder
Brief Title: Carvedilol Versus Placebo for Treatment in Post Traumatic Stress Disorder (PTSD)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Columbia Northwest Pharmaceuticals (Industry)
Responsible Party: Arifulla Khan, MD, Columbia Northwest Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CVD-PT-10203
Record Dates: First submitted 2010-10-14; First posted 2010-10-15 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-06

CONDITIONS: Post-Traumatic Stress Disorder
Keywords: PTSD; Anxiety; Trauma; Assault; Victim; Witness; Post Traumatic Stress Disorder; Combat veteran; Flashbacks; Nightmares; Sleep Disturbance; Hyperarousal; Numbness; Avoidance
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Anxiety Disorders; Wounds and Injuries; Parasomnias; Hypesthesia | interventions — Carvedilol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- carvedilol (Active Comparator): Patients randomized to carvedilol will be administered doses ranging from 6.25 to 15.625 mg/day using a flexible-dosing model. After a 1 week titration, investigators my increase daily dose by 6.25 mg/day at weeks 1 and 2 for a maximum dose of 15.625 mg/day. Weeks 3-4 will patients will remain on a stable, tolerable dose. At week 5 patients will have a 1 week taper.
  Interventions: Drug: Carvedilol
- Sugar Pill (Placebo Comparator): Patients randomized to placebo will follow same dosing guidelines as if they were in the active comparator arm, carvedilol.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Carvedilol — Oral, twice daily dosing using 3.125 mg tablets.
  1 week titration (6.25 mg/day)prior to a 3 week flexible dosing option ranging from 6.25 mg/day to 15.625 mg/day followed by a 1 week taper (6.25 mg/day).
  Other Names: Coreg(R)
  Arms: carvedilol
Drug: Placebo — Non active comparator
  Arms: Sugar Pill

SUMMARY:
The investigators hypothesize that carvedilol, at less then therapeutic doses for cardiac effect, will reduce symptoms of Post Traumatic Stress Disorder.

DETAILED DESCRIPTION:
This initial proof of concept trial design is intended to explore multiple variables. Fist, it is intended to determine if carvedilol has any statistically significant effect over placebo on the various overall symptoms, symptom clusters, or individual symptoms of post traumatic stress disorder. Next, the flexible dosing trial design is aimed to detect the therapeutic dose, or dosing range for carvedilol when used in the treatment of PTSD

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Post Traumatic Stress Disorder according to DSM-IV
* Must be able to speak, read and understand the English language and be able to provide written informed consent

Exclusion Criteria:

* current, unstable and significant medical condition/illness
* bronchial asthma or related bronchospastic condition
* AV block
* Sick Sinus Syndrome
* Bradycardia
* Peripheral hear disease
* Unstable thyroid disorder
* History of seizure disorder
* Females who are pregnant, lactating or planning to become pregnant
* Bipolar
* Schizophrenia
* Dementia
* Intolerance or hypersensitivity to alpha or beta blockers

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2010-10; Primary Completion 2011-06 (Estimated); Study Completion 2011-08 (Estimated)

PRIMARY OUTCOMES:
Davidson Trauma Scale (DTS) | 5 weeks
  The DTS is a 17-item self report measure to assess the 17 DMS-IV symptoms of PTSD. Respondants are asked to identify the trauma that is most disturbing to them and to rate, in the past week, how much trouble they hav had with each symptom. The DTS can be used to make a preliminatry determination about whether the symptoms meet DSM criteria for PTSD, or scores can be calculated for each of the 3 PTSD symptom clusters.
  The DTS will be assessed at each study visit (visit 1, 2, 3, 4, 5, 6 and 7). The primary efficacy outcome will be change from baseline (visit 2) to week 5 (visit 7).

SECONDARY OUTCOMES:
Clinician Administered PTSD Scale (CAPS) | 6 Weeks
  The CAPS was developed at the National Center for PTSD and has become the "gold standard" for assessing Post Traumatic Stress Disorder. It is a user-friendly structured interview for screening, differential diagnosis, comfirming PTSD diagnosis or identifying Acute Stress Disorder.
  The CAPS will be assessed at the screening visit and again at week 5 (vist 7). Change scores (from screening to week 5) will be secondary efficacy measures.
Insomnia Severity Index (ISI) | 5 Weeks
  The ISI is a 7-item patient rated questionnaire that evaluates severity of sleep onset and maintenance difficulties, satisfaction with current sleep pattern interference with daily functioning, appearance of impairment attributed to the sleep problem, and the degree of concern caused by insomnia.
  Secondary outcome measures using the ISI will be determined using change scores from baseline to week 5 (visit 7)

CONTACTS AND LOCATIONS:
Overall Officials: Arifulla Khan, MD, Study Director — Columbia Northwest Pharmaceuticals, LLC
Locations (3):
- United States (3):
  - Artemis Institute for Clinical Research, San Diego, California
  - Lake Charles Clinical Trials, Lake Charles, Louisiana
  - Northwest Clinical Research Center, Bellevue, Washington